CLINICAL TRIAL: NCT00213577
Title: Evaluation of the Efficacy and Tolerance of 2 Dosages of Type A Botulinic Toxin in Neurogenic Areactive Bladder Resistant to Oral Medical Treatment
Brief Title: NEUROTOX: Two Dosages of Type A Botulinic Toxin in Neurogenic Overactive Bladder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the study has concluded normally;
Sponsor: University Hospital, Rouen (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2003/112/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Overactive Bladder
Keywords: overactive neurogenic bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: type A botulinum toxin

SUMMARY:
The purpose of this study is to determine the efficacy and tolerance of 2 dosages (750 versus 500 units) of the Dysport type A botulinic toxin for patient suffering from neurogenic urinary incontinence by an overactive bladder and the failure of anticholinergic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Neurogenic urinary incontinence with urodynamic overactivity resistant to anticholinergic

Exclusion Criteria:

* Pregnancy
* Bladder cancer
* Symptomatic urinary infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-12; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
complete urinary continence at baseline, and days 30, 90, 180, and 360

SECONDARY OUTCOMES:
number of mictions or self catheterizations a day
number of leakages, urgency adverse events
guarding times
urodynamics: bladder capacity, reflex volume, residual maximal capacity detrusor pressure, flow detrusor pressure

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GRISE, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- CHU-Rouen, Rouen, France

REFERENCES:
- [Derived] Grise P, Ruffion A, Denys P, Egon G, Chartier Kastler E. Efficacy and tolerability of botulinum toxin type A in patients with neurogenic detrusor overactivity and without concomitant anticholinergic therapy: comparison of two doses. Eur Urol. 2010 Nov;58(5):759-66. doi: 10.1016/j.eururo.2010.06.035. Epub 2010 Jul 3. PMID 20674149